CLINICAL TRIAL: NCT02251015
Title: Evaluation of Postural Balance in Individuals With Temporomandibular Disorder by Means of Force Platform After Using Occlusal Stabilizer Splint Disorder
Brief Title: Effects of the Use of Occlusal Splint on the Postural Balance of Individuals With Temporomandibular Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Simone Saldanha Ignacio de Oliveira, Effects of the use of occlusal splint on the postural balance of individuals with temporomandibular disorder, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Postural balance
Record Dates: First submitted 2013-11-06; First posted 2014-09-26 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Temporomandibular Disorders
Keywords: Postural balance; Temporomandibular disorders; splints
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- therapeutic exercises (Active Comparator): 13 as control group - The control group got only orientation related to therapeutic exercises.The orientation for therapeutic exercises seek to correctly position the jaw in the resting position. Maxillary teeth approximately 2mm away from the mandibular teeth and the tip of the tongue accommodated on top of the incisive papilla on the hard palate, beyond an exercise that consisted of repeated opening and closing movements paying close attention to the position of the tongue, the point of which being accommodated on the incisive papilla during the exercises. The patient was instructed to perform 15 repetitions 3 times a day.
  Interventions: Procedure: therapeutic exercises
- occlusal plate group (Experimental): 36 getting occlusal splints - the splinted group was subjects that used occlusal plate under the occlusal stability criteria. The patients also received therapeutic exercises too. The plate group arm, the patients used the occlusal splints for all night plus 4 hours during the day and they made therapeutic exercises 15 repetitions 3 times a day.
  Interventions: Procedure: occlusal plate; Procedure: therapeutic exercises

INTERVENTIONS:
Procedure: occlusal plate — In the plate group arm, the patients used the occlusal splints for all night plus 4 hours during the day and they made therapeutic exercises 15 repetitions 3 times a day.
  The orientation for therapeutic exercises seek to correctly position the jaw in the resting position (maxillary teeth approximately 2mm away from the mandibular teeth and the tip of the tongue accommodated on top of the incisive papilla on the hard palate, beyond an exercise that consisted of repeated opening and closing movements paying close attention to the position of the tongue, the point of which being accommodated on the incisive papilla during the exercises. The patient was instructed to perform 15 repetitions 3 times a day.
  Arms: occlusal plate group
Procedure: therapeutic exercises — The orientation for therapeutic exercises seek to correctly position the jaw in the resting position (maxillary teeth approximately 2mm away from the mandibular teeth and the tip of the tongue accommodated on top of the incisive papilla on the hard palate, beyond an exercise that consisted of repeated opening and closing movements paying close attention to the position of the tongue, the point of which being accommodated on the incisive papilla during the exercises. The patient was instructed to perform 15 repetitions 3 times a day.

SUMMARY:
To investigate the effects of the use of occlusal splint over postural balance in individuals with signs and symptoms of temporomandibular disorder. The research group consists of 49 patients (36 getting occlusal splints and 13 as control group) between 18 and 75 years old, both genders, diagnosed as temporomandibular disorder (TMD) by RDC/TMD questionnaire and magnetic resonance imaging of the temporomandibular joints. The research is a randomized, controlled, prospective clinical study with intervention. Postural equilibrium will be evaluated by means of a force plate. In the randomization, the splinted group was under an occlusal-stability criterion as well as advised under therapeutic exercises while the control group got only orientation about therapeutic exercises. After 12 weeks, the groups were re-evaluated. The results will be analyzed by categorical data using absolute and relative frequencies as well as continuous data using average, median, standard deviation, 25 and 75 percentiles, besides minimum and maximum values; comparison between the times by non-parametric Wilcoxon, Mann-Whitney and ANOVA tests with a threshold of significance of 0.05.

DETAILED DESCRIPTION:
approved 06/29/2011

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic Criteria Temporomandibular Disorders and dentate subjects

Exclusion Criteria:

* Without Diagnostic Criteria Temporomandibular Disorders and edentulous subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
to investigate the effects of the use of occlusal splint over postural balance in individuals with signs and symptoms of temporomandibular disorder. | twelve weeks
  Postural equilibrium was evaluated by means of a force plate. In the randomization, the splinted group was under an occlusal-stability criterion as well as advised under therapeutic exercises while the control group got only orientation related to therapeutic exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Simone de Oliveira, PHD, Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo/SP, Brazil